CLINICAL TRIAL: NCT03594435
Title: A Randomized Controlled Clinical Trial of the Neuroimmune Modulator Ibudilast for the Treatment of Alcohol Use Disorder
Brief Title: Ibudilast for the Treatment of Alcohol Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); MediciNova (Industry)
Responsible Party: Principal Investigator, Lara Ray, PhD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-000963; R01AA026190 (NIH)
Record Dates: First submitted 2018-07-11; First posted 2018-07-20 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Alcohol Use Disorder
Keywords: ibudilast, treatment, medication development
MeSH Terms: conditions — Alcoholism | interventions — ibudilast; Sugars

STUDY DESIGN:
Intervention Model Description: Two-Arm, Randomized, Double-Blind, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ibudilast (Experimental): 10mg delayed-release capsules, target dose 50mg twice daily (5 x 10mg capsules twice daily) for 12 weeks
  Interventions: Drug: Ibudilast
- Placebo Oral Capsule (Placebo Comparator): matched to experimental drug
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Ibudilast — targets neurotrophin signaling and neuroimmune function
  Other Names: Pinatos; MN-166
  Arms: Ibudilast
Drug: Placebo oral capsule — matched to active drug, ibudilast
  Other Names: Sugar Pill
  Arms: Placebo Oral Capsule

SUMMARY:
This study is a double-blind, placebo-controlled randomized clinical trial of Ibudilast (IBUD) (50mg twice a day) for the treatment of Alcohol Use Disorder (AUD). Eligible participants will undergo a 12-week medication treatment period and 5 in-person visits over 16 weeks.

DETAILED DESCRIPTION:
The study design consists of a 12-week, double-blind, placebo-controlled randomized clinical trial of IBUD (50mg twice a day) for the treatment of AUD. The investigators will randomize 132 treatment-seekers with current AUD over the course of 4 years. Participants will complete telephone screening, followed by in-person eligibility assessment, a physical exam for medical eligibility, randomization to study medication or matched placebo, and in-person follow-up visits at 4, 8, and 12 weeks of treatment. Timeline Followback (TLFB) assessment of drinking outcomes will also occur by telephone on weeks 2, 6, and 10. A final safety check visit will occur on week 16, consisting of repeated clinical labs and electrocardiography (ECG).

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 18 and 65
2. Meet current (i.e., past 12 months) Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) diagnostic criteria for alcohol use disorder moderate or severe
3. Be treatment-seeking for alcohol use disorder (AUD)
4. Report drinking at least 28 drinks per week if male (21 drinks per week if female) in the 28 days prior to consent

Exclusion Criteria:

1. Have a current (last 12 months) DSM-5 diagnosis of substance use disorder for any psychoactive substances other than alcohol and nicotine
2. Have a lifetime DSM-5 diagnosis of schizophrenia, bipolar disorder, or any psychotic disorder
3. Have a positive urine screen for narcotics, amphetamines, or sedative hypnotics;
4. Have clinically significant alcohol withdrawal symptoms as indicated by a score ≥ 10 on the Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-R)
5. Be pregnant, nursing, or planning to become pregnant while taking part in the study; and must agree to one of the following methods of birth control (if female), unless she or partner are surgically sterile:

   * Oral contraceptives
   * Contraceptive sponge
   * Patch
   * Double barrier
   * Intrauterine contraceptive device
   * Etonogestrel implant
   * Medroxyprogesterone acetate contraceptive injection
   * Complete abstinence from sexual intercourse
   * Hormonal vaginal contraceptive ring
6. Have a medical condition that may interfere with safe study participation (e.g., unstable cardiac, renal, or liver disease, uncontrolled hypertension or diabetes)
7. Have aspartate aminotransferase (AST), alanine transaminase (ALT), or gamma-glutamyl transferase (GGT) ≥ 3 times upper normal limit
8. Have attempted suicide in the past 3 years and/or have had serious suicidal intention or plan in the past year
9. Currently be on prescription medication that contraindicates use of ibudilast (IBUD), including alpha or beta agonists, theophylline, or other sympathomimetic
10. Currently be on any medications for AUD or any psychotropic medications (e.g., psychostimulants and benzodiazepines) with the exception of stable antidepressants (stable dose for ≥4 weeks)
11. Have any other circumstances that, in the opinion of the investigators, compromises participant safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lara A. Ray, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Addictions Laboratory, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McManus KR, Enders C, Kirsch DE, Belnap M, Grodin EN, Ray LA. Peripheral inflammation mediates the relationship between early life stress and alcohol use. Psychopharmacology (Berl). 2026 Jan 28. doi: 10.1007/s00213-026-07009-8. Online ahead of print. PMID 41603979
- [Derived] Ray LA, Meredith LR, Grodin EN, Belnap MA, Nieto SJ, Baskerville WA, Donato S, Shoptaw SJ, Gillis AJ, Irwin MR, Miotto K, Enders CK. A Neuroimmune Modulator for Alcohol Use Disorder: A Randomized Clinical Trial. JAMA Netw Open. 2025 Apr 1;8(4):e257523. doi: 10.1001/jamanetworkopen.2025.7523. PMID 40305022
- [Derived] Burnette EM, Baskerville WA, Grodin EN, Ray LA. Ibudilast for alcohol use disorder: study protocol for a phase II randomized clinical trial. Trials. 2020 Sep 11;21(1):779. doi: 10.1186/s13063-020-04670-y. PMID 32912290

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via online and print advertisements, local bus campaigns, and targeted recruitment through a laboratory database of previous study participants who agreed to be contacted for further studies.
Pre-assignment Details: A stratified randomization list was developed by a statistician and was based on gender, drinking status (moderate drinking defined as ≥ 14 drinks/week for men and ≥ 7 drinks/week for women versus heavy drinking defined as ≥ 28 drinks/week for men and ≥ 21 drinks/week for women).
Groups:
- Ibudilast: 10mg delayed-release capsules, target dose 50mg twice daily (5 x 10mg capsules twice daily) for 12 weeks
  ibudilast: targets neurotrophine signaling and neuroimmune function
Period: Overall Study
Arm/Group | Ibudilast | Placebo Oral Capsule
Started | 53 | 49
Completed | 48 | 41
Not Completed | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibudilast | Placebo Oral Capsule | Total
Number analyzed (Participants) | 53 | 49 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.74 (10.01) | 45.92 (11.49) | 44.26 (10.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 32 | 29 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 16 | 32
  Not Hispanic or Latino | 37 | 33 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 13 | 11 | 24
  White | 25 | 27 | 52
  More than one race | 7 | 6 | 13
  Unknown or Not Reported | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 53 | 49 | 102
Drinks per drinking day [Mean (Standard Deviation); unit: drinks per drinking day] — Drinks per drinking day at baseline was measured using the timeline followback. This measure is defined as the number of drinks a participant had on a reported day of drinking during the 30-day prior to the baseline visit.
  drinks per drinking day | 7.57 (4.30) | 7.52 (3.36) | 7.54 (5.36)
Percent heavy drinking days [Mean (Standard Deviation); unit: percent heavy drinking days] | 67.5 (34.55) | 65.7 (34.89) | 66.6 (34.55)
Number of drinking days [Mean (Standard Deviation); unit: drinking days] | 22.42 (7.46) | 22.71 (7.41) | 22.56 (7.40)
Positive THC screen [Count of Participants; unit: Participants] | 23 | 11 | 34
Mild Cannabis Use Disorder [Count of Participants; unit: Participants] | 6 | 6 | 12
Any cigarette use [Count of Participants; unit: Participants] — Any cigarette use as indexed by any reported cigarette use on the past 30-day timeline followback.
  Participants | 18 | 17 | 35
Smokes cigarettes [Count of Participants; unit: Participants] — Smokes cigarettes was measured using item 1 of the Fagerstrom Test for Nicotine Dependence ('How often do you smoke (cigarettes)?'). Participants who marked daily or occasionally were identified as participants who smoke cigarettes and those who marked not at all were identified as participants who do not smoke cigarettes.
  Participants | 20 | 20 | 40
Penn Alcohol Craving Scale Total [Mean (Standard Deviation); unit: units on a scale] — The Penn Alcohol Craving Scale (PACS) measures alcohol craving. The total score ranges from 0 to 30 with higher scores indicating more alcohol craving.
  units on a scale | 13.83 (5.85) | 13.73 (6.56) | 13.78 (6.17)
Structured Clinical Interview Alcohol Use Disorder symptom count [Mean (Standard Deviation); unit: units on a scale] — The Structured Clinical Interview of Alcohol Use Disorder (AUD) symptom count measures the number of AUD symptoms participants endorse. Symptom count ranges from 0 to 11, with 0-1 symptoms indicating no alcohol disorder, 2-3 symptoms indicating mild alcohol use disorder, 4-5 symptoms indicating moderate alcohol use disorder, and 6 or more symptoms indicating severe alcohol use disorder.
  units on a scale | 7.15 (2.05) | 6.27 (1.69) | 6.73 (1.93)
Alcohol Use Disorders Identification Test [Mean (Standard Deviation); unit: units on a scale] — The Alcohol Use Disorder Identification Test (AUDIT) identifies individuals with hazardous and harmful patterns of alcohol consumption. Total scores range from 0 to 40. A score of 1-7 indicates low risk consumption, scores 8-14 indicate hazardous or harmful alcohol consumption, and 15 or more indicates likelihood of alcohol dependence.
  units on a scale | 21.23 (8.24) | 19.16 (6.14) | 20.24 (7.35)
Relief/Habit Drinking [Count of Participants; unit: Participants] | 27 | 25 | 52
Current Depression [Count of Participants; unit: Participants] | 4 | 3 | 7
Beck's Depression Inventory-II Total [Mean (Standard Deviation); unit: units on a scale] — The Beck's Depression Inventory-II (BDI-II) captures depressive symptomatology. Total scores range from 0 to 63. Scores between 0-9 indicates minimal depression, 10-18 indicates mild depression, 19-29 indicates moderate depression, and 30-63 indicates severe depression.
  units on a scale | 11.98 (8.55) | 10.73 (7.13) | 11.38 (7.89)
Beck's Anxiety Inventory Total [Mean (Standard Deviation); unit: units on a scale] — The Beck's Anxiety Inventory (BAI) measures anxiety symptomatology including physical and cognitive indicators of anxious mood. Total scores range from 0 to 63. A score between 0-7 indicates minimal anxiety, 8-15 indicates mild anxiety, 16-25 indicates moderate anxiety, and 26-63 indicates severe anxiety.
  units on a scale | 8.53 (7.87) | 6.94 (7.08) | 7.76 (7.51)
Insomnia Severity Index Total [Mean (Standard Deviation); unit: units on a scale] — The Insomnia Severity Index (ISI) assess symptoms of insomnia. Total scores range from 0-28. Scores between 0-7 indicate no clinical significant insomnia, 8-14 indicates sub-threshold insomnia, 15-21 indicates clinical insomnia (moderately severity), and 22-28 indicates clinical insomnia (severe).
  units on a scale | 9 (6.29) | 7.98 (5.23) | 8.51 (5.80)

OUTCOME MEASURES:

1. Primary Outcome: Percent Heavy Drinking Days
Description: Heavy drinking days defined as 5+ drinks for men and 4+ for women. Reported outcome measures are proportions of heavy drinking days.
Time Frame: 12 week-treatment period
Measure: Mean (Standard Deviation); unit: percent of heavy drinking days
Arm/Group | Ibudilast | Placebo Oral Capsule
Number analyzed (Participants) | 53 | 49
percent of heavy drinking days
  Randomization | 67.4777 (34.54664) | 65.65447 (34.89305)
  Week 2 Follow-up | 53.88376 (38.62032) | 42.96028 (42.12516)
  Week 4 Follow-up | 48.57848 (40.24403) | 43.54836 (42.40074)
  Week 6 Follow-up | 40.13970 (41.51441) | 45.83959 (39.41569)
  Week 8 Follow-up | 47.88029 (40.47520) | 35.80680 (40.36051)
  Week 10 Follow-up | 43.36704 (40.82088) | 37.54797 (40.80282)
  Week 12 Follow-up | 34.96705 (38.75223) | 35.33841 (40.07343)

2. Secondary Outcome: Drinks Per Day
Description: Secondary alcohol consumption endpoint. Outcome measure reported is the proportion of drinks per day. Drinks per day across the trial. Randomization is the first day of study intervention after study eligibility was determined.
Time Frame: 12-week treatment period
Measure: Mean (Standard Deviation); unit: Drinking per day
Groups:
- Ibudilast: 10mg delayed-release capsules, target dose 50mg twice daily (5x 10mg capsules twice daily) for 12 weeks
  ibudilast: targets neurotrophin signaling and neuroimmune function
Arm/Group | Ibudilast | Placebo Oral Capsule
Number analyzed (Participants) | 53 | 49
Drinking per day
  Randomization | 5.5569643 (3.8825400) | 5.0916392 (3.2844504)
  Week 2 Follow-up | 2.9712639 (2.6163298) | 2.5307298 (2.5759514)
  Week 4 Follow-up | 2.9416414 (3.0687885) | 2.7376672 (2.2163207)
  Week 6 Follow-up | 2.9004471 (3.1327782) | 2.4886257 (1.9787647)
  Week 8 Follow-up | 2.5295239 (2.0967361) | 1.9764896 (2.0375665)
  Week 10 Follow-up | 2.3335342 (2.2920357) | 1.9942146 (1.9999379)
  Week 12 Follow-up | 2.2639331 (2.2143404) | 1.9131006 (2.0874590)

3. Secondary Outcome: Drinks Per Drinking Day
Description: Secondary alcohol consumption endpoint. Drinks per drinking day is defined as how many drinks an individual consumed on a day they reported drinking alcohol.
Time Frame: 12-week treatment period
Measure: Mean (Standard Deviation); unit: drinks per drinking day
Arm/Group | Ibudilast | Placebo Oral Capsule
Number analyzed (Participants) | 53 | 49
drinks per drinking day
  Randomization | 7.5702563 (4.3026834) | 7.5157381 (6.3591036)
  Week 2 Follow-up | 6.0380129 (4.2269696) | 4.6825232 (3.6986878)
  Week 4 Follow-up | 5.1232947 (3.6194523) | 4.8648040 (4.2417622)
  Week 6 Follow-up | 4.8955457 (3.9859161) | 4.4555121 (3.1474673)
  Week 8 Follow-up | 4.9961214 (3.4733168) | 3.4954873 (2.7084074)
  Week 10 Follow-up | 4.6825531 (4.1278832) | 3.3946192 (2.5414040)
  Week 12 Follow-up | 4.1250715 (3.1777328) | 3.4113607 (2.4958175)

4. Secondary Outcome: Percent Days Abstinent
Description: Secondary alcohol consumption endpoint. Outcome measure reported is the proportion of percent days abstinent.
Time Frame: 12-week treatment period
Measure: Mean (Standard Deviation); unit: percent days abstinent.
Arm/Group | Ibudilast | Placebo Oral Capsule
Number analyzed (Participants) | 53 | 49
percent days abstinent.
  Randomization | 25.28269 (24.86230) | 24.28538 (24.71130)
  Week 2 Follow-up | 52.10013 (31.53534) | 51.24152 (36.33756)
  Week 4 Follow-up | 53.49783 (33.79115) | 46.76799 (35.31845)
  Week 6 Follow-up | 50.14506 (34.61062) | 49.30242 (36.06276)
  Week 8 Follow-up | 49.85351 (35.34000) | 54.99929 (38.86134)
  Week 10 Follow-up | 56.10048 (34.49246) | 54.35469 (37.55533)
  Week 12 Follow-up | 54.86251 (34.42088) | 55.35643 (38.60974)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participant between randomization to Week 12 visit (final day of study).
Description: The study physician (Dr. Miotto) called every participant at the end of the first week on the study medication to discuss any adverse events. Adverse events were also collected at each monthly visit and the study physician was notified of any reported adverse events.
Arm/Group | Ibudilast | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/49
Serious Adverse Events (participants affected / at risk) | 1/53 | 1/49
Other Adverse Events (participants affected / at risk) | 36/53 | 27/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibudilast (N=53) | Placebo Oral Capsule (N=49)
Left Upper Quadrant Abdominal Pain (General disorders) | 0 | 1
Left Ankle Open Fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural Hematoma (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibudilast (N=53) | Placebo Oral Capsule (N=49)
Insomnia (General disorders) | 4 | 3
Anxiety (Psychiatric disorders) | 4 | 4
Diarrhea (Gastrointestinal disorders) | 4 | 2
Vomiting (Gastrointestinal disorders) | 5 | 3
Headache (General disorders) | 8 | 8
Flu like symptoms (General disorders) | 4 | 4
Body pain (General disorders) | 8 | 6
Nausea (Gastrointestinal disorders) | 8 | 8
Fatigue (General disorders) | 4 | 1
Dizziness (General disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 2
Depression (Psychiatric disorders) | 2 | 2
Libido (Reproductive system and breast disorders) | 0 | 1
Gut pain (Gastrointestinal disorders) | 3 | 4
Skin discoloration (Skin and subcutaneous tissue disorders) | 0 | 1
Dysmenorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 3
Sweating (General disorders) | 1 | 2
Flushing (General disorders) | 1 | 0
Hypertension (Blood and lymphatic system disorders) | 1 | 0
Abnormal EKG (Cardiac disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Blurry vision (Eye disorders) | 1 | 2
Pain and discomfort (General disorders) | 11 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT03594435/Prot_SAP_000.pdf